CLINICAL TRIAL: NCT04909723
Title: Phase 1-2a Safety, Tolerability, and Pharmacodynamics Controlled Study of NOV-001 in Healthy Volunteers and Patients With Enteric Hyperoxaluria
Brief Title: Safety, Tolerability, and Pharmacodynamics of NOV-001 in Adult Subjects
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision to discontinue study.
Sponsor: Novome Biotechnologies Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NOV-001-CL01
Record Dates: First submitted 2021-05-07; First posted 2021-06-02 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Healthy Volunteers; Enteric Hyperoxaluria
Keywords: Healthy volunteers; Safety; Tolerability; Enteric hyperoxaluria; Kidney stone; Roux-en-Y gastric bypass; Hyperoxaluria; Secondary hyperoxaluria; Oxalate; Kidney calcification; Gastric bypass; Biliopancreatic diversion with duodenal switch; Duodenal switch
MeSH Terms: conditions — Kidney Calculi; Hyperoxaluria

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Stage 1 placebo arm (Placebo Comparator)
  Interventions: Drug: Placebo
- Stage 1 NB1000S 10^9 CFU one time on Day 1 (Experimental)
  Interventions: Biological: NB1000S
- Stage 1 NB1000S 10^9 CFU one time on Day 1 and NB2000P 0.5g/day (Experimental)
  Interventions: Combination Product: NOV-001
- Stage 1 NB1000S 10^9 CFU one time on Day 1 and NB2000P 10g/day (Experimental)
  Interventions: Combination Product: NOV-001
- (Optional) Stage 1 variable doses of NB1000S and NB2000P at varying dosing regimens. (Experimental): Adaptive trial design supports the enrollment of additional arms with variable doses of NB1000S, NB2000P, at varying frequencies of NB1000S and NB2000P administrations.
  Interventions: Combination Product: NOV-001
- Stage 1 NB2000P at a dose to be determined (Experimental)
  Interventions: Drug: NB2000P
- Stage 2 NOV-001 at dose determined in Stage 1 (Experimental): In Stage 2, subjects will be randomized (3:1, NOV-001:placebo) to receive NOV-001 (consisting of NB1000S and NB2000P at a dose and regimen determined in Stage 1) for 28 days.
  Interventions: Combination Product: NOV-001
- Stage 2 placebo arm (Placebo Comparator): In Stage 2, subjects will be randomized (3:1, NOV-001:placebo) to receive placebo for 28 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Combination Product: NOV-001 — NOV-001 is an investigational combination product composed of NB1000S, a recombinant live biotherapeutic product, and NB2000P, a botanically derived polysaccharide.
  Arms: (Optional) Stage 1 variable doses of NB1000S and NB2000P at varying dosing regimens.; Stage 1 NB1000S 10^9 CFU one time on Day 1 and NB2000P 0.5g/day; Stage 1 NB1000S 10^9 CFU one time on Day 1 and NB2000P 10g/day; Stage 2 NOV-001 at dose determined in Stage 1
Biological: NB1000S — A recombinant live biotherapeutic product.
  Arms: Stage 1 NB1000S 10^9 CFU one time on Day 1
Drug: NB2000P — A botanically derived polysaccharide.
  Arms: Stage 1 NB2000P at a dose to be determined
Drug: Placebo — Placebo
  Arms: Stage 1 placebo arm; Stage 2 placebo arm

SUMMARY:
The first stage of this study is a prospective, adaptive, Phase 1, first-in-human, randomized, controlled study evaluating safety, tolerability, and pharmacodynamics of NOV-001 in adult healthy volunteers.

The second stage of this study is a prospective, randomized, single-blinded, placebo-controlled study of safety, tolerability, and early efficacy in patients with enteric hyperoxaluria.

DETAILED DESCRIPTION:
This study is evaluating the safety, tolerability, pharmacodynamics, and early efficacy of NOV-001. NOV-001 is an investigational combination product composed of NB1000S, a recombinant live biotherapeutic product, and NB2000P, a botanically derived polysaccharide. In Stage 1, NB1000S (or placebo) is administered on the first day of treatment and NB2000P is administered once daily, or as indicated in the adaptive study design. In Stage 2, NB1000S (or placebo) is administered two times per day on the first day of the treatment and NB2000P (or placebo) is administered once daily for 28 days, at doses determined in Stage 1.

ELIGIBILITY:
Stage 1 Key Inclusion Criteria:

* Ages 18 to 55
* Body mass index (BMI) < 38 kg/m2.
* Healthy as defined by no clinically relevant abnormalities being identified by a detailed medical history, physical examination, and clinical laboratory tests.
* If woman of child-bearing potential, must not be pregnant, and must also agree to use an appropriate highly-effective contraceptive.
* Willing and able to comply with all study requirements, including duration of stay at inpatient unit, dietary restrictions, daily study product administration, pregnancy testing and contraception (if applicable), stool collections, and blood and urine collections.

Stage 1 Key Exclusion Criteria:

* Estimated glomerular filtration rate (eGFR) < 80 mL/min/1.73 m2 at Screening.
* Oral or parenteral antibiotics within 4 weeks prior to Screening, or anticipation of the need for such antibiotics during the Screening or treatment periods of the study.
* Current or history of any clinically significant medical illness or disorder the Investigator considers should exclude the subject from the study.
* Participation in any investigational intervention study within 30 days prior to study product administration in this study.
* Known hypersensitivity to omeprazole.
* Applicable only to certain study groups depending on emerging Stage 1 data: no current or anticipated use during the screening or treatment periods of the study of medications that have the potential for drug-drug interactions (DDI) with omeprazole.

Stage 2 Key Inclusion Criteria:

* Ages 18 to 65.
* Hyperoxaluria secondary to Roux-en-Y gastric bypass surgery or to biliopancreatic diversion with duodenal switch (BPD-DS) surgery.
* 24-Hour urinary oxalate (UOx) ≥ 60 mg.
* If woman of child-bearing potential, must not be pregnant and must also agree to use an appropriate highly effective contraceptive method.
* Must, in the opinion of the Investigator, be in otherwise good health.
* Willing and able to comply with all study requirements, including dietary restrictions, daily study product administration, pregnancy testing and contraception (if applicable), stool collections, and blood and 24-hour urine collections.

Stage 2 Key Exclusion Criteria:

* Chronic kidney disease with eGFR < 30 mL/min/1.73 m2 at Screening.
* Evidence of current acute renal injury or ongoing clinically significant renal disease.
* Oral or parenteral antibiotics within 4 weeks prior to Screening, or anticipation of the need for such antibiotics during the Screening or treatment periods of the study (topical antibiotics are permissible.)
* Taking during the study any treatment for hyperoxaluria except for NOV-001, other than stable treatments for the management of kidney stones.
* Taking Vitamin C ≥ 300 mg/day for > 10 days within 7 days prior to Screening; unwilling or unable to discontinue and/or avoid Vitamin C supplementation for the duration of study product treatment.
* Known active autoimmune disorder or other condition requiring high dose of systemic corticosteroids (i.e., > 10 mg/day prednisone or equivalent) or other immunosuppressant therapy.
* Current or history of any clinically significant medical illness or disorder other than enteric hyperoxaluria that the Investigator considers should exclude the patient from the study.
* Participation in any investigational intervention study within 30 days prior to study product administration in this study.
* Known hypersensitivity to omeprazole.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v5.0 | Up to 182 days

OTHER OUTCOMES:
NB1000S engraftment as measured by quantitative Polymerase Chain Reaction (qPCR) determination of concentration of NB1000S strain genomic copies (cells/mL) in stool, change from baseline. | Up to 182 days
The proportion of subjects with NB100S strain abundance in stool, as measured by qPCR determination of concentration of strain genomic copies (cells/mL). | Up to 182 days
Time to strain engraftment, based on the time to reach NB1000S strain abundance by qPCR determination of concentration of NB1000S strain genomic copies (cells/mL). | Up to 182 days
Fecal shedding of NB1000S strain as measured by qPCR determination of concentration of NB1000S strain genomic copies (cells/mL), during treatment and follow-up periods. | Up to 182 days
Absolute change from baseline in 24-hour urinary oxalate (UOx) excretion (mg/mL), NOV-001 compared to placebo. | Stage 2; 28 days
Percent change from baseline in 24-hour UOx excretion (mg/mL), NOV-001 compared to placebo. | Stage 2; 28 days
Proportion of patients achieving ≥ 20% reduction in 24-hour UOx excretion from baseline to end of treatment, NOV-001 compared to placebo. | Stage 2; 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Lachy McLean, MB ChB, PhD, Study Director — Novome Biotechnologies Inc
Locations (20):
- United States (19):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic, Scottsdale, Arizona
  - Advanced Urology Institute, Daytona Beach, Florida
  - Prohealth Research Center, Doral, Florida
  - Florida Urology Partners, Tampa, Florida
  - Georgia Clinical Research, Lawrenceville, Georgia
  - Idaho Urologic Institute, Meridian, Idaho
  - Indiana University, Carmel, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Chesapeake Urology Associates, Hanover, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St. Louis, St Louis, Missouri
  - Associated Urologists of North Carolina, Raleigh, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Clinical Research Solutions, Cleveland, Ohio
  - The Miriam Hospital, Providence, Rhode Island
  - AMR Knoxville, Knoxville, Tennessee
  - Knoxville Kidney Center, Knoxville, Tennessee
  - Houston Metro Urology, Houston, Texas
- Alpha Recherche Clinique, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No